CLINICAL TRIAL: NCT05580120
Title: The Effect of an Online-supervised Exercise Program in Elderly People With Diabetes on Fasting Blood Sugar, Psychological Resilience, and Quality of Life: A Double Blind Randomize Controlled Trial
Brief Title: Online-supervised Exercise Program in Elderly People With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Ersoy University (Other)
Collaborators: Akdeniz University (Other)
Responsible Party: Principal Investigator, Nurten Terkes, Principal Investigator, Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GO 2021/293
Record Dates: First submitted 2022-10-07; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Exercise Program; Type2diabetes
Keywords: psychological resilience; quality of life; distance education

STUDY DESIGN:
Who Masked: Participant
Masking Description: They did not know if they were in the control and intervention group at the time of randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online-supervised exercise group (Experimental): After the pre-tests (The Brief Resilience Scale, Quality of Life) , the patients were given online-supervised exercise education for 6 weeks.
  Interventions: Behavioral: Online-supervised exercise group
- The unsupervised-exercise training group (Experimental): After the pre-tests (The Brief Resilience Scale, Quality of Life) , the patients were given unsupervised exercise education for 6 weeks.
  Interventions: Behavioral: Unsupervised-exercise training group

INTERVENTIONS:
Behavioral: Online-supervised exercise group — Participants in the online-supervised exercise group were provided with an online-supervised exercise program by using the video conferencing method three times a week for 6 weeks on the Zoom application. The exercise program was carried out synchronously
  Arms: Online-supervised exercise group
Behavioral: Unsupervised-exercise training group — The unsupervised-exercise training group was informed about how to do the same exercises by another researcher, a nurse academician, on the online platform by using the lecturing method. Each training intervention took approximately 30 minutes.
  Arms: The unsupervised-exercise training group

SUMMARY:
This study was conducted to determine the effect of an online-supervised exercise program on fasting blood sugar, psychological resilience, and quality of life in elderly people with diabetes. A parallel-group, randomized controlled trial design was used. The study was conducted in a public hospital with 70 patients with elderly type 2 diabetes between Nowember 2021 and May 2022. A Personal Information Form, The Brief Resilience Scale and A Measure of Quality of Life in the Elderly were used to collect data.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of Type 2 diabetes mellitus for at least 6 months,
* Being aged >50 years,
* Receiving oral antidiabetic and/or insulin therapy,
* Having a smartphone or a computer,
* Volunteering to participate in the study,

Exclusion Criteria:

* Individuals who had type 2 DM, but were illiterate
* Had vision and hearing loss
* Did not volunteer to participate in the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
The Brief Resilience Scale | 5 minute
  The scale was developed by Smith et al. to measure individuals' resilience levels and was adapted to Turkish by Doğan. It is a one-dimensional 6-item measurement tool. High scores obtained from the scale indicate that the individual's psychological resilience is good. Cronbach's alpha internal consistency coefficient of the scale is .83.
A Measure of Quality of Life in the Elderly | 5 minute
  This scale was developed by Hyde et al. in 2003 to measure the quality of life of the elderly. It was adapted to Turkish society in 2014 by Türkoğlu and Adıbelli. An increase in the total score indicates an increase in the quality of life. The scale consists of two sub-dimensions, namely "perceived autonomy and satisfaction" and "perceived disability". Cronbach's alpha value of the original scale is .91.

CONTACTS AND LOCATIONS:
Overall Officials: Sabriye Ucan Yamac, PhD, Study Chair — Burdur Mehmet Akif Ersoy University
Locations (1):
- Burdur Mehmet Akif Ersoy University, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All authors contributed to the interpretation, writing, and approval of the final manuscript.

REFERENCES:
- [Result] Ruiz-Roso MB, Knott-Torcal C, Matilla-Escalante DC, Garcimartin A, Sampedro-Nunez MA, Davalos A, Marazuela M. COVID-19 Lockdown and Changes of the Dietary Pattern and Physical Activity Habits in a Cohort of Patients with Type 2 Diabetes Mellitus. Nutrients. 2020 Aug 4;12(8):2327. doi: 10.3390/nu12082327. PMID 32759636
- [Result] Duruturk N, Ozkoslu MA. Effect of tele-rehabilitation on glucose control, exercise capacity, physical fitness, muscle strength and psychosocial status in patients with type 2 diabetes: A double blind randomized controlled trial. Prim Care Diabetes. 2019 Dec;13(6):542-548. doi: 10.1016/j.pcd.2019.03.007. Epub 2019 Apr 20. PMID 31014938
- [Result] Seron P, Oliveros MJ, Gutierrez-Arias R, Fuentes-Aspe R, Torres-Castro RC, Merino-Osorio C, Nahuelhual P, Inostroza J, Jalil Y, Solano R, Marzuca-Nassr GN, Aguilera-Eguia R, Lavados-Romo P, Soto-Rodriguez FJ, Sabelle C, Villarroel-Silva G, Gomolan P, Huaiquilaf S, Sanchez P. Effectiveness of Telerehabilitation in Physical Therapy: A Rapid Overview. Phys Ther. 2021 Jun 1;101(6):pzab053. doi: 10.1093/ptj/pzab053. PMID 33561280